CLINICAL TRIAL: NCT00682461
Title: A Randomized, Open Label Study to Evaluate the Oral Tolerability of a Nicotine Prototype
Brief Title: Oral Tolerability Of Two Nicotine Dosage Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2110367
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Volunteer Smokers
Keywords: Nicotine Tolerability NRT
MeSH Terms: interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marketed formulation (Active Comparator): Marketed nicotine replacement therapy product
  Interventions: Drug: Nicotine
- prototype (Experimental): Nicotine prototype
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Marketed nicotine replacement therapy formulation
  Other Names: marketed NRT formulation
  Arms: Marketed formulation
Drug: Nicotine — Nicotine prototype
  Other Names: Nicotine prototype
  Arms: prototype

SUMMARY:
This study is to evaluate the oral tolerability of a nicotine prototype

ELIGIBILITY:
Inclusion Criteria:

* Age:Males and females aged at least 18 years.
* Smoking status: a.Must have smoked 5 to 20 cigarettes per day for the previous 12 months. b.Must be motivated to quit smoking upon randomization into study.
* Contraception:Females of childbearing potential who have been, in the opinion of the investigator, practicing a reliable method of contraception for at least two months prior to study participation and must agree to remain on an acceptable method of contraception while participating in the study period using the study medication. Acceptable methods of contraception are hormonal birth control, intrauterine device, double barrier methods, vasectomized partner or abstinence.
* Oral health:Must have good oral health (in the opinion of the Investigator) with no clinically significant oral pathology at screening.
* General health:Must have good general health (in the opinion of the Investigator) with no clinically significant and relevant abnormalities of medical history on physical examination at screening.
* Compliance:Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Consent:Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.

Exclusion Criteria:

* Pregnancy:Women who are known to be pregnant or who are intending to become pregnant over the duration of the study. Females of child-bearing potential will be required to undergo a urine pregnancy test which must be negative.
* Breast-feeding:Women who are breast-feeding.
* Nicotine use: a.Is unable/unwilling to stop using forms of tobacco. b.Is unable/unwilling to stop using other nicotine replacement therapy.
* Disease:Has a medical history, which in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results, e.g. known history of heart disease, recent myocardial infarction or cerebrovascular accident (i.e. within 12 weeks prior to the first study session), unstable angina, severe cardiac arrhythmia, diabetes or peptic ulcer.
* Oral condition: a.Has history of oral surgery (including extractions) within four weeks, operative dental work within seven days, or a presence of any clinically significant oral pathology (as determined by the Investigator) including lesions, sores or inflammation which would interfere with assessments. b.Has fixed retainers, orthodontic appliances, or either maxillary and/or mandibular dentures or other appliances which may interfere with the placement or wearing of the product. c.Has current or recurrent disease that could affect the site of application, the action, absorption or disposition of the study treatment, or clinical assessment. d.Has severe gingivitis, periodontitis or rampant caries, as diagnosed by the investigator. e.Has the presence of oral or peri-oral ulceration including herpetic lesions at the time of baseline (subjects with these lesions may be re-examined at a subsequent appointment and may be able to be admitted at a later date if the ulceration or herpetic lesion heals). f.Has elective dentistry scheduled during the study duration.
* Allergy/Intolerance: a.Has a known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients. b.Presence of a genetic deficiency with an inability to metabolize aspartame or phenylalanine or has been diagnosed with phenylketonuria.
* Clinical Study/Experimental medication: a.Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit at the start of the study. b.Previous participation in this study.
* Substance abuse: a) Current or recent (within two year of screening) alcohol or other substance abuse. b) Positive alcohol breath screen. c) Positive urine drug screen for cannabinoids, amphetamine, cocaine, ecstasy, methamphetamine or morphine.
* Urine glucose:Positive glucose urine screen.
* Personnel: a.Is an employee of the sponsor or the study site. b.Is a member of the same household as another subject in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one clinical site in the US.
Groups:
- Nicotine Mouth Strip (2.5 mg): Participants were instructed to take 2.5 mg Nicotine Mouth Strip, not exceeding a maximum limit of 15 per day
- Nicotine Lozenge (2.0 mg): Prticipants were instructed to take 2.0 mg Nicotine Lozenge, not exceeding a maximum limit of 15 per day
Period: Overall Study
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Started | 100 | 100
Completed | 75 | 69
Not Completed | 25 | 31
Not completed — Adverse Event | 5 | 7
Not completed — Lost to Follow-up | 8 | 5
Not completed — Withdrawal by Subject | 12 | 19

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Lozenge (2.0 mg): Participants were instructed to take 2.0 mg Nicotine Lozenge, not exceeding a maximum limit of 15 per day
- Total: Total of all reporting groups
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.32 (11.79) | 42.84 (12.34) | 42.58 (12.042)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 63 | 125
  Male | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Oral Soft Tissue Related Adverse Events at Week 1
Description: Oral Soft Tissue related adverse events= Any abnormality occuring in any of these: labial mucosa (including lips), gingival mucosa, buccal mucosa, mucogingival folds, hard and soft palates, tonsilar and pharyngeal areas, tongue, sublingual and submandibular areas, and salivary glands
Time Frame: From baseline to Week 1
Population: Analysis was based on safety population, which consisted of all randomized participants who took at least one dose of the study medication.
Measure: Number; unit: Percentage
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Number analyzed (Participants) | 86 | 87
Percentage | 2.3 | 12.6

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Adverse Event=any untoward medical occurrence in a subject following administration of an investigational product, which did not necessarily have a causal relationship with this treatment.
  Serious Adverse Event=any untoward medical occurrence that at any dose; results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect
Time Frame: From baseline to Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Number analyzed (Participants) | 100 | 100
Percentage
  Oral Treatment Emergent Adverse Events | 27 | 44
  Non-oral Treatment Emergent Adverse Events | 58 | 60
  Serious Adverse Events | 0 | 1
  Death | 0 | 0

3. Primary Outcome: Percentage of Participants With Oral Soft Tissue Related Adverse Events at Week 6
Description: as for outcome 1
Time Frame: From baseline to Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Number analyzed (Participants) | 76 | 73
Percentage | 6.6 | 12.3

4. Primary Outcome: Percentage of Participants With Oral Soft Tissue Related Adverse Events at Week 12
Description: as for outcome 1
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Number analyzed (Participants) | 75 | 70
Percentage | 6.7 | 7.1

5. Primary Outcome: Percentage of Participants With Oral Soft Tissue Related Adverse Events at Week 14
Description: as for outcome 1
Time Frame: From baseline to Week 14
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Number analyzed (Participants) | 82 | 87
Percentage | 2.4 | 8.0

ADVERSE EVENTS:
Time Frame: From baseline to Week 14
Description: All adverse events
Groups:
- Nicotine Lozenge (2.0 mg): Participants were instructed to take 2.0 mg Nicotine Lozenge, not exceeding a maximum of 15 per day
Arm/Group | Nicotine Mouth Strip (2.5 mg) | Nicotine Lozenge (2.0 mg)
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/100
Other Adverse Events (participants affected / at risk) | 69/100 | 75/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Mouth Strip (2.5 mg) (N=100) | Nicotine Lozenge (2.0 mg) (N=100)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Unrelated to the study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Mouth Strip (2.5 mg) (N=100) | Nicotine Lozenge (2.0 mg) (N=100)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 13 (15)
Mouth Injury (Injury, poisoning and procedural complications) | 5 (5) | 6 (8)
Oral Mucosal Erythema (Gastrointestinal disorders) | 1 (2) | 3 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Tooth Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival Ulceration (Gastrointestinal disorders) | 1 (1) | 3 (4)
Oral Discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 11 (12) | 14 (17)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 8 (8)
Flatulence (Gastrointestinal disorders) | 0 (0) | 7 (7)
Gastrointestinal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooenteritis Viral (Infections and infestations) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 17 (18) | 19 (20)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 9 (11) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.